CLINICAL TRIAL: NCT05913258
Title: Evaluation of Caries Removal in Primary Teeth Using an Er:YAG Laser: A Randomized Split-Mouth Clinical Trial
Brief Title: Caries Removal in Primary Teeth Using Er:YAG Laser
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: King Abdulaziz University (Other)
Responsible Party: Principal Investigator, Osama M Felemban, Associate Professor in Pediatric Dentistry, King Abdulaziz University
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: KAUFD Er:YAG 20230525
Record Dates: First submitted 2023-05-25; First posted 2023-06-22 (Actual); Last update posted 2023-06-22 (Actual); Status verified 2023-06

CONDITIONS: Dental Caries
MeSH Terms: conditions — Dental Caries

STUDY DESIGN:
Intervention Model Description: A randomized, blinded split-mouth study. The children were randomly assigned into one of two groups randomly. The first group included were assigned to receive the conventional treatment at the first visit and the laser treatment at the second visit. The second group was assigned to receive the laser treatment at the first visit and the conventional treatment at the second visit.
Who Masked: Outcomes Assessor
Masking Description: The examiner who clinically evaluated the restorations using Ryge criteria did not know which tooth had received which treatment.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Er:YAG Laser Caries Removal group (Experimental): Complete isolation was performed using a rubber dam and saliva ejector. Patients received topical anesthesia before the clamp was placed. Dental caries was excavated using the Er:YAG laser with a wavelength of 2940nm according to the manufacturer's instructions until visual inspection showed that the carious lesions have been thoroughly removed. If the patient experienced pain and requested local anaesthesia, the procedure was stopped, local anaesthesia has been applied, and then the procedure has resumed. Cavities were restored using the Clearfil Universal Bond Quick system in total each mode; 37% phosphoric acid was used, then the Clearfil Universal Bond system was applied, light cured for 90 seconds, after which composite resin was applied (3M Filtek TM Z350 XT Universal Restorative Composite (3M ESPE) according to the manufacturer's instructions.
  Interventions: Device: Er:YAG laser system (Doctor smile, Pluser, Italy)
- Conventional Caries Removal Group (Active Comparator): Complete isolation was performed using a rubber dam and saliva ejector. Patients received topical anesthesia before the clamp was placed. Dental caries was excavated using the Mastertorque high/low-speed air rotor handpiece until visual inspection showed that the carious lesions have been thoroughly removed. If the patient experienced pain and requested LA, the procedure was stopped, LA was applied, and then the procedure resumed. According to the manufacturer's instructions, cavities were restored using the Clearfil Universal Bond Quick system and composite resin (3M Filtek TM Z350 XT Universal Restorative Composite (3M ESPE).
  Interventions: Device: Master Torque high/low-speed air rotor handpiece (KaVo Dental, Charlotte, North Carolina, USA)

INTERVENTIONS:
Device: Er:YAG laser system (Doctor smile, Pluser, Italy) — The Er:YAG laser offers a virtually painless alternative to conventional methods of caries removal, and its adoption in clinical practice could greatly reduce children's fear of going to the dentist. Caries removal is one of the leading reasons for dentist visits among children, and many children become fearful at the mere thought of a drill touching their teeth, before they even hear the sound. Laser caries removal could go a long way toward eliminating children's fear of going to the dentist; it is virtually painless, and most children are able to get through the entire procedure without needing local anesthesia.
  Arms: Er:YAG Laser Caries Removal group
Device: Master Torque high/low-speed air rotor handpiece (KaVo Dental, Charlotte, North Carolina, USA) — Mechanical removal of carious lesions with a rotating handpiece and bur instruments is the most often used approach for treating dental caries because it is cost-effective, timesaving, and simple. However, these procedures have many drawbacks, including the potential for removing healthy tooth structures, vibration and noise, which can cause the patient anxiety and pain, thus necessitating local anesthesia.
  Arms: Conventional Caries Removal Group

SUMMARY:
Objective: To assess and compare the 2940 nm erbium:yttrium-aluminum-garnet (Er:YAG) laser versus a conventional rotary treatment during cavity preparation in children with regard to anxiety level, pain perception, restoration integrity, and bond interface quality.

Materials and Methods: In a randomized, blinded trial using a split-mouth design, forty (9-12-year-old) children with 80 carious deciduous molars were included. The cavity in one quadrant was treated conventionally using a bur, while the cavity in the other quadrant was prepared using an Er:YAG laser. Venham's dental anxiety scale and pulse rate measurement using a fingertip pulse oximeter were used to evaluate dental anxiety levels. The Wong-Baker facial pain rating scale and the number of local anesthesia required during both interventions were further applied to investigate pain perception. At the 1-year follow-up, clinical examinations was conducted and the integrity of the restorations was clinically assessed according to the Ryge criteria. Lastly, the restored teeth were extracted and histologically evaluated for bond interface quality using scanning electronic microscopy.

DETAILED DESCRIPTION:
Study Design: A randomized, blinded split-mouth study was conducted with a sample of 40 healthy children aged 9 to 12 years (N=40 children) / (n=80 teeth). The children were divided into two groups randomly. The first group included 20 children who were assigned to receive the conventional treatment at the first visit and the laser treatment at the second visit (N=20 children) / (n=40 teeth). The second group was assigned to receive the laser treatment at the first visit and the conventional treatment at the second visit (N=20 children) / (n=40 teeth). Both groups received the laser and conventional treatment and were assessed for pain and anxiety during both interventions. After a follow -up period of 1 year, an analysis of the restorative integrity evaluation was performed using the Ryge criteria. The restored teeth were extracted according to the normal exfoliation schedule and analyzed for bond interface quality evaluation.

Study Sample: Study participants were recruited from the patient population at the pediatric dentistry clinics at King Abdulaziz University Dental Hospital in Jeddah, Saudi Arabia. Every patient in the appropriate age range has been examined for class I carious lesions of the molars, and in patients where these molars were present, the researcher was notified by the practitioner. The researcher was to make the final decision about the suitability of patients to be included in the study sample. The researcher explained the study procedures to the parents of potential subjects, and if they agreed to participate, consent to participate in the study has been obtained from the parents of the pediatric patients.

Sample Size Calculation: According to the authors' assumptions, a sample size of 31 pairs will have 80 percent power to detect a difference in proportions of restorations integrity of 0.2 when the proportion of discordant pairs is expected to be 0.21, and the analysis method is a McNemar's test of equality of paired proportions with a 5% two-sided significance level.

Randomization Procedure: Each patient has undergone conventional caries removal on one affected molar and laser caries removal on the other. The researcher prepared 80 sealed envelopes divided into two groups in 2 boxes, each containing 40 envelopes. The first group was for the treatment procedures randomization, 20 of which contained instructions to perform conventional caries removal on the first tooth and laser caries removal on the second, and other 20 contained instructions to use the laser on the first tooth and the rotary bur on the second. The second group for tooth randomization consisted of 40 envelopes, 20 of which contained instructions to treat the tooth in the right quadrant first, and 20 of which contained instructions to treat the tooth in the left quadrant first. The envelopes were identical from the outside, only the messages inside differed. The subjects, who did not know the contents of the envelopes, were asked to select two envelopes, one from each group. The researcher opened them and read the contents to be informed as to which treatment and which tooth would be performed first.

Treatment Procedure: The conventional treatment and the laser treatment took place at two separate visits, approximately one week apart, with the order of the treatments to be determined by the randomization process. The teeth were restored using Clearfil Universal Bond Quick self-etching primer, bonding resin and Clearfil APX composite resin.

One-Year-Follow-Up: Follow-up took place one year later, at which time clinical examination was conducted. The integrity of the restorations has been clinically examined. The examiner did not know which tooth had received which treatment. The restorations were evaluated according to Ryge criteria; the criteria published by the United States Public Health Service. The criteria that were measured included: anatomical form, axial contour, marginal contact, margin discoloration, secondary caries, and visible plaque. Each criterion received a numerical rating from zero to two (zero to three for some criteria) and a score of Alpha, Bravo, or Charlie (or Delta for marginal contact and axial contour.

Teeth Extractions: The restored teeth were followed up for two more years and were extracted whenever it was determined that the root of the successor's tooth was formed (according to the normal tooth shedding time of the patient). The extracted teeth were evaluated for bond interface quality.

ELIGIBILITY:
Inclusion Criteria:

* Healthy patients between 9 and 12 years of age.
* Simple occlusal caries that is limited to enamel and dentine without proximal caries, or pulp involvement in at least two primary molars (pairs).
* Primary molars with 1/3rd of their root remained.
* Primary teeth have permanent successor teeth with 1/2 of the root formed.

Exclusion Criteria:

* Caries lesion that had reached or was approaching the pulp.
* Previous fillings.
* Periapical lesions, or dental abscess.
* No permanent successor teeth.
* Behavioral or medical problem.

Ages: 9 Years to 12 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 40 (Actual)
Dates: Start 2020-01-01 (Actual); Primary Completion 2022-03-01 (Actual); Study Completion 2022-03-01 (Actual)

PRIMARY OUTCOMES:
Venham's Behavior Rating Scale (VBRS). | The treatment procedure (which lasted about 30-45 minutes) was video recorded from start to end. Later, two observers watched the videos to assign each subject a score reflecting his/her behavior throughout the whole procedure time from start to end.
  Venham's Behavior Rating Scale is an interval rating scale in which the rating procedure is reliable, valid, and can be easily integrated into clinical or research activities. It is a six-point scale, ranging from 0 to 5 with scale points anchored in objective, specific, and readily observable behavior. Higher scores indicate higher anxiety.
Baseline Heart rate. | The baseline heart rate reading was recorded at the beginning of the dental visit immediately after the subject sat on the dental chair.
  Heart rate measurement is a direct measure of physiological arousal since its increase is attributed to stress during dental procedures. A pulse oximeter was used to measure the heart rate. The pulse oximeter was placed on the subject finger at the beginning of the dental visit immediately after he/she sat on the dental chair and remained in place until the treatment was completed.
Mean Heart rate. | The mean heart rate was calculated by averaging the heart readings recorded every 5 minutes from the start until the end of the dental procedure.
  Heart rate measurement is a direct measure of physiological arousal since its increase is attributed to stress during dental procedures. A pulse oximeter was used to measure the heart rate. The pulse oximeter was placed on the subject finger at the beginning of the dental visit immediately after he/she sat on the dental chair and remained in place until the treatment was completed. Heart rate readings were recorded every 5 minutes until the treatment procedure was finished which lasted about 30-45 minutes.
Wong-Baker Pain Scale | Immediately after the caries excavation procedure was done, subjects were asked to choose the face on the Wong-Baker Faces Pain Rating Scale that best depicts the pain they were experiencing during treatment.
  The Wong-Baker scale is a pictorial scale appropriate for children three years and older, that uses pictures of different facial expressions representing different levels of pain from 0-10, face 0 doesn't hurt at all, face 2 hurts just a little bit, face 4 hurts little bit more, face hurts even more, face 8 hurt a whole lot, face 10 hurts as much as you can imagine.
Local Anesthesia Administration | The injection of local anesthesia anytime during the 30 to 45 minute dental visit.
  During the dental procedure, if the child experienced pain and requested local anesthesia, the procedure was stopped, local anesthesia was injected, and then the procedure resumed. The number of children who requested local anesthesia during any of the interventions, conventional or laser, was documented.

SECONDARY OUTCOMES:
Restorations' Integrity Evaluation | follow-up visit one year after the restorations were placed.
  The restorations were evaluated according to Ryge criteria. The criteria that were measured included: anatomical form, axial contour, marginal contact, margin discoloration, secondary caries, and visible plaque. Each criterion received a numerical rating from zero to three and a score of Alpha, Bravo, or Charlie or Delta.

CONTACTS AND LOCATIONS:
Locations (1):
- King Abdulaziz University, Jeddah, Saudi Arabia